CLINICAL TRIAL: NCT00848315
Title: Diabetes Management in Low-Income Hispanic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R18DK065985 (NIH)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes; Glycemic Control
Keywords: cognitive behavioral intervention; low literate/illiterate Hispanic patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual Care that the Type 2 Diabetes Patients usually receive at the health centers.
- 2 (Experimental): Cognitive Behavioral Intervention
  Interventions: Behavioral: Cognitive Behavioral Intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Intervention — The intervention emphasizes patients' ethnic preferences and traditions (e.g., adapting ethnic recipes to meet dietary goals) and the use of available community resources (e.g., available areas for exercise), and is delivered utilizing strategies and materials appropriate for low-literate/illiterate patients.
  Other Names: Diabetes Self-Management
  Arms: 2

SUMMARY:
The overall goal of this randomized clinical trial (RCT) is to test the efficacy of a culturally- and literacy-tailored cognitive-behavioral intervention designed to enhance adherence to diabetes self-management behaviors and improve glycemic control among low-income Hispanic individuals with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Patients are randomly assigned to a Usual Care condition or to the Cognitive Behavioral Intervention condition. The unit of randomization and analysis is the patient. The intervention is implemented by a nutritionist, a nurse diabetes educator and an assistant, and patients are encouraged to bring a family member or friend living in the same household to facilitate home-based support for the intervention. The intervention emphasizes patients' ethnic preferences and traditions (e.g., adapting ethnic recipes to meet dietary goals) and the use of available community resources (e.g., available areas for exercise), and is delivered utilizing strategies and materials appropriate for low-literate/illiterate pts.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with T2DM (documented in the medical chart);
2. HbA1c level > 7.5;
3. Currently treated with diet, oral hypoglycemics or insulin. If currently on insulin, must have a history of prior therapy with diet alone or oral hypoglycemic agents;
4. Hispanic origin;
5. > 18 years old;
6. Telephone in home or easy access to one;
7. Able to understand and participate in the study protocol;
8. Functionally capable of meeting the activity goals;
9. Understands and can provide informed consent (English or Spanish; for illiterate pts we will require that a representative of the pt also understands and signs the consent form on behalf of the pt);
10. Physician approval to participate in the study.

Exclusion Criteria:

1. History of diabetic ketoacidosis
2. Gestational diabetes
3. Unable or unwilling to provide informed consent;
4. Plans to move out of the area within the 12-month study period;
5. Required intermittent glucocorticoid therapy within the past 3 months;
6. Experienced an acute coronary event (myocardial infarction or unstable angina) within the previous 6 mos
7. Has a medical condition that precludes adherence to study dietary recommendations (e.g., Crohn's disease, ulcerative colitis, end-stage renal disease);
8. Has a medical or psychiatric illness (i.e., dementia, psychiatric hospitalization or suicidality within past 5 years or takes an atypical neuroleptic medication). We will not exclude individuals with a diagnosis of depression or pts taking anti-depressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is improvement in metabolic control (HbA1c). | The primary outcome was evaluated at 4- and 12-months following randomization.

SECONDARY OUTCOMES:
Efficacy of the intervention | 4- and 12-months following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Milagros C Rosal, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (5):
- United States (5):
  - Northgate Medical Center, Springfield, Massachusetts
  - Brightwood Health Center, Springfield, Massachusetts
  - High Street Health Center, Springfield, Massachusetts
  - Plumley Village, Worcester, Massachusetts
  - Family Health Center, Worcester, Massachusetts

REFERENCES:
- [Derived] Wang ML, Gellar L, Nathanson BH, Pbert L, Ma Y, Ockene I, Rosal MC. Decrease in Glycemic Index Associated with Improved Glycemic Control among Latinos with Type 2 Diabetes. J Acad Nutr Diet. 2015 Jun;115(6):898-906. doi: 10.1016/j.jand.2014.10.012. Epub 2014 Dec 26. PMID 25547339
- [Derived] Rosal MC, White MJ, Restrepo A, Olendzki B, Scavron J, Sinagra E, Ockene IS, Thompson M, Lemon SC, Candib LM, Reed G. Design and methods for a randomized clinical trial of a diabetes self-management intervention for low-income Latinos: Latinos en Control. BMC Med Res Methodol. 2009 Dec 9;9:81. doi: 10.1186/1471-2288-9-81. PMID 20003208